CLINICAL TRIAL: NCT00727012
Title: Multicenter International Trial Ring AnnulopLasty
Acronym: MITRAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Prof. Dr. Raffaele De Simone, University of Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS06003RG
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Mitral Valve Insufficiency
Keywords: mitral valve; heart valve; valve repair; valve disorder; valve disease; cardiac surgery
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SJM® Rigid Saddle Ring (Other): The SJM® Rigid Saddle Ring is an annuloplasty ring comprised of a titanium core surrounded by a double-velour, polyester fabric sewing cuff.
  Interventions: Device: mitral valve repair (SJM® Rigid Saddle Ring)

INTERVENTIONS:
Device: mitral valve repair (SJM® Rigid Saddle Ring) — mitral valve repair due to mitral degenerative or functional disease

SUMMARY:
This clinical study is a multicenter, prospective non-randomized observational study without concurrent or matched controls in which 150 patients receiving an SJM® Rigid Saddle Ring will be included. The primary objective of the study is to demonstrate the effectiveness of the SJM® Rigid Saddle Ring when used in mitral valve repair procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a mitral valve repair due to mitral degenerative or functional disease (Note: Patients that underwent concomitant procedures, e.g. coronary artery bypass grafting, are eligible for this study);
* Patient (or legal guardian) has signed a study specific informed consent form agreeing to the data collection and follow-up requirements;
* Patients are at least 18 years old.

Exclusion Criteria:

* Patient requires replacement of the aortic, tricuspid or pulmonary valve or has a pre-existing prosthetic valve;
* Patient is pregnant or nursing;
* Patient has active endocarditis;
* Patient is actively participating in another study of an investigational drug or device;
* Patients unavailable to follow-up visit (abroad residents, patients affected by neurological disorders...);
* Patients who are intravenous drug abusers, alcohol abusers, prison inmates or unable to give informed consent;
* Patients with a major non-cardiac evolving disease;
* Patients with a life expectancy less than 1 year;
* Patients are known to be noncompliant or are unlikely to complete the study;
* Any case in which mitral annuloplasty rings are not indicated;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in ERO (Effective Regurgitant Orifice) in cm2 calculated with PISA method at 6 months and at patient discharge compared to baseline (pre-operative). | 6 months
NYHA class | 6 months

SECONDARY OUTCOMES:
adverse events rates | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Simone, Prof. Dr., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany